CLINICAL TRIAL: NCT02101892
Title: Prediction of Migraine Prevention Efficacy: Individualization of Treatment by Coupling Drug's Mode of Action With Patient's Mechanism of Pain Modulation
Brief Title: Prediction of Migraine Prevention Efficacy Based on Individual's Pain Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Migraine Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0102-14
Record Dates: First submitted 2014-03-18; First posted 2014-04-02 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Migraine; Preventive Treatment
Keywords: migraine; Amitriptyline; pain modulation; pain psychophysics; pain neurophysiology; preventive treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amitriptyline (Active Comparator): Amitriptyline, 25 mg per os, daily, evening, for 8 weeks; starting dose is 12.5 mg for 2 days
  Interventions: Drug: placebo
- placebo (Placebo Comparator): sugar pills
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — per os, daily, evening
  Other Names: Elatrol
  Arms: placebo
Drug: placebo — per os, daily, evening
  Other Names: sugar pills
  Arms: Amitriptyline

SUMMARY:
A major reason for the substantial underuse of pharmacological prevention of migraine is its inadequate efficacy, since only ~50% of patients respond to a specific agent. There is currently no evidence-based way to identify the patients that will respond to a specific preventive treatment. Amitriptyline is one of the commonest agents used for migraine prevention, strengthening patient's pain inhibitory capacity. Individual tailoring of analgesics according to pain inhibitory capacity has been shown effective by our group for painful diabetic neuropathy patients. Specifically, patients with reduced pain inhibition capacity gained more from a drug that augment pain inhibition as compared to those with efficient inhibitory capacity. The investigators now propose to assess migraineurs for their pain inhibition capacity, and examine whether, along similar reasoning, those with reduced inhibitory capacity are the ones more likely to respond to amitriptyline. Psychophysical and neurophysiological dimensions of pain inhibitory modulation will be assessed in migraineurs, who will, subsequently, receive either amitriptyline or placebo for 8 weeks, in a randomized two arms parallel double blind design, and followed up for attacks reduction. The investigators expect to identify the best predictors for efficacy of migraine prevention by the study drug. This approach will promote individualization of migraine therapy.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* premenopausal
* meeting the international headache society criteria for migraine
* having >4 attacks or days of migraine/month

Exclusion Criteria:

* baseline month diary indicating lower frequency of migraine
* chronic migraine (>15 days of headache per month)
* use of migraine preventive treatment during previous 3 month
* language barrier or cognitive dysfunction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
predictive value of the pre-treatment pain measures parameter(s) for benefit from amitriptyline treatment | one year
  ANCOVA will be utilized, based on factors treatment (amitriptyline or placebo), conditioned pain modulation capabilities (responder or non-responder), their interaction, a number of covariates, to predict reduction attacks.

SECONDARY OUTCOMES:
predictive value of pain-related psychological parameters for benefit from amitriptyline treatment | one year
  The scores for Spielberger's anxiety state and trait questionnaire, and for pain catastrophising questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, MD, Professor, Principal Investigator — Rambam Health Care Campus and Technion Medical School; Yelena Granovsky, PhD, Principal Investigator — Rambam Health Care Campus and Technion Medical School; Michal Granot, Professor, Principal Investigator — Nursing School, University of Haifa
Locations (1):
- Rambam Health Care Campus, Haifa, Israel